CLINICAL TRIAL: NCT02759809
Title: Optimizing Mothers' Milk for Preterm Infants (OptiMoM) Program of Research: Study 1-Impact of Donor Milk at Kindergarten
Brief Title: OptiMoM Kindergarten Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, Research Institute, The Hospital for Sick Children
Other Study IDs: 1000053053
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Infant, Very Low Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Children previously assigned to donor milk in the DoMINO trial: This study is an observational study of children who were enrolled in a previous trial (DoMINO trial) between 2010 and 2012 during which they were randomized to receive donor milk when mother's own breastmilk was unavailable. Donor milk was from a milk bank part of the Human Milk Banking Association of North America (HMBANA).
  Interventions: Other: Pasteurized donor human breastmilk
- Children previously assigned to formula in the DoMINO trial: This study is an observational study of children who were enrolled in a previous trial (DoMINO trial) between 2010 and 2012 during which they were randomized to receive preterm formula when mother's own breastmilk was unavailable. Preterm formula was either Similac Special Care or Enfamil Premature depending on hospital contract with formula companies.
  Interventions: Other: Preterm formula

INTERVENTIONS:
Other: Pasteurized donor human breastmilk
  Groups: Children previously assigned to donor milk in the DoMINO trial
Other: Preterm formula
  Groups: Children previously assigned to formula in the DoMINO trial

SUMMARY:
In Canada, the leading cause of long-term disability in children is being born at very low birth weight (VLBW). To help improve outcomes, nutrition is a modifiable aspect of infant care. Mother's milk is the optimal way to feed VLBW infants; however, many need a supplement of donor milk or preterm formula as not enough mother's milk is available. As the ideal supplement for prolonged feeding and its long-term effects is currently unknown, this study is a prospective follow up of VLBW infants who in hospital were fed: donor milk or preterm formula and/or mother's milk. Areas of development to be assessed include: cognition, language, motor skills, brain structure/function, and body composition. A DNA biorepository will also be created.

ELIGIBILITY:
Inclusion Criteria:

* Children who were enrolled in the DoMINO (Donor Milk for Improved Neurodevelopmental Outcomes) trial (ISRCTN35317141).

Ages: 5 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Very low birth weight infants previously enrolled in the DoMINO (Donor Milk for Improved Neurodevelopmental Outcomes) trial (ISRCTN35317141).
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Full-Scale IQ on the Wechsler Preschool and Primary Scale of Intelligence-IV (WPPSI-IV) | 5.5 years of age

SECONDARY OUTCOMES:
Verbal IQ on the WPPSI-IV | 5.5 years of age
Performance IQ on the WPPSI-IV | 5.5 years of age
General Language Composite on the WPPSI-IV | 5.5 years of age
Processing Speed Quotient on the WPPSI-IV | 5.5 years of age
Growth | 5.5 years of age
  Growth as assessed using weight, height and waist circumference measurements.
Body Composition | 5.5 years of age
  Body composition as assessed using the COSMED BOD POD and skinfold thickness.

OTHER OUTCOMES:
Affect Recognition domain on the NEPSY-II | 5.5 years of age
Language domain on the NEPSY-II | 5.5 years of age
Memory domain on the NEPSY-II | 5.5 years of age
Visual-Motor Integration using the Beery | 5.5 years of age
Development of Brain Structure | 5.5 years of age
  Development of brain structure as assessed using Magnetic Resonance Imaging (MRI).
Development of Brain Function | 5.5 years of age
  Development of brain function as assessed using Magnetoencephalography (MEG).
Interaction of genetic differences and feeding type on outcomes | 5.5 years of age
  Assessed using a buccal cell biorepository.
Influence of the diet on epigenetic changes | 5.5 years of age
  Assessed using a buccal cell biorepository.
School Readiness using the Early Development Instrument (EDI) | 5.5 years of age

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Xu J, Shin J, McGee M, Unger S, Bando N, Sato J, Vandewouw M, Patel Y, Branson HM, Paus T, Pausova Z, O'Connor DL. Intake of mother's milk by very-low-birth-weight infants and variation in DNA methylation of genes involved in neurodevelopment at 5.5 years of age. Am J Clin Nutr. 2022 Oct 6;116(4):1038-1048. doi: 10.1093/ajcn/nqac221. PMID 35977396
- [Derived] Walton K, McGee M, Sato J, Law N, Hopperton KE, Bando N, Kiss A, Unger SL, O'Connor DL. Social-emotional functioning and dietary intake among children born with a very low birth weight. Appl Physiol Nutr Metab. 2022 Jul 1;47(7):737-748. doi: 10.1139/apnm-2021-0434. Epub 2022 Feb 23. PMID 35196153
- [Derived] McGee M, Unger S, Hamilton J, Birken CS, Pausova Z, Kiss A, Bando N, O'Connor DL. Associations between Diet Quality and Body Composition in Young Children Born with Very Low Body Weight. J Nutr. 2020 Nov 19;150(11):2961-2968. doi: 10.1093/jn/nxaa281. PMID 33025010
- [Derived] McGee M, Unger S, Hamilton J, Birken CS, Pausova Z, Kiss A, Bando N, O'Connor DL. Adiposity and Fat-Free Mass of Children Born with Very Low Birth Weight Do Not Differ in Children Fed Supplemental Donor Milk Compared with Those Fed Preterm Formula. J Nutr. 2020 Feb 1;150(2):331-339. doi: 10.1093/jn/nxz234. PMID 31599955
- See also: Donor Milk for Improved Neurodevelopmental Outcomes (DoMINO) trial — http://www.controlled-trials.com/ISRCTN35317141